CLINICAL TRIAL: NCT05710419
Title: Effects of Invasive Mechanical Ventilation on the Right Ventricular Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: 157/22
Record Dates: First submitted 2023-01-03; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Pneumonia; Atelectasis; ARDS
MeSH Terms: conditions — Pneumonia; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the influence of mechanical ventilation on the right ventricular (RV) function. The primary focus is on methods which are routinely used to improve gas exchange in ventilated patients (positive end expiratory pressure [PEEP], inhalation of NO, prone positioning). The main questions it aims to answer are:

* Effects of prone positioning, PEEP and inhalation of NO on RV-function
* Are there determinants (clinical, laboratory, demographic, echocardiographic) for the right ventricular response to the above?

RV-Function will be assessed with right ventricular pressure-volume loops recorded with a conductance catheter at

* each PEEP-Level during titration of the best PEEP
* before and every 5 minutes (for max. 45 minutes) after rotation to prone position
* before and under continuous inhalation of NO (if required based on clinical grounds)

DETAILED DESCRIPTION:
Pressure-volume loop (PV-loop) analysis is the gold standard for the assessment of right ventricular properties and function in clinical research. PV-Loops can be generated in real-time by conductance catheterization, which allows a simultaneous acquisition of pressure and volume changes in high resolution. It is known that invasive mechanical ventilation, primarily through a change in intrathoracic pressure conditions, has a significant impact on the function of the right ventricle. However, the underlying mechanisms have not yet been investigated and understood in detail using the gold standard. Therefore, the aim of this observational study is to investigate the effects of invasive ventilation and ventilatory strategies to improve gas exchange (PEEP, prone position, inhaled NO) on the function of the right ventricle.

The physiology of mechanical ventilation is fundamentally different than spontaneous breathing: While in spontaneous breathing the air fills the lungs driven by a negative intrathoracic pressure, in mechanical ventilation air has to be "pumped" into the lungs, resulting in a positive intrathoracic pressure. These unphysiological intrathoracic pressure conditions lead to complex interactions between the respiratory and cardiovascular system, can stress the right ventricle and cause hemodynamic instability. In addition to the stress of mechanical ventilation per se, there are changes in the pulmonary vasculature in caused by the pulmonary disease itself. A maximum expression of such changes is the acute respiratory failure syndrome (ARDS), which requires a complex ventilation strategy and is associated with a high mortality rate. ARDS is always associated with a dysfunction of the pulmonary vessels (hypoxic vasoconstriction, pulmonary microthrombosis, derecruitment of ventilated areas) leading to increased right ventricular afterload. In contrast to the left ventricle, the right ventricle has only a small contractile reserve and is therefore more sensible to a higher afterload. This is why the right ventricle can be seen as the weakest link of the circulatory system in patients with ARDS. This is also reflected in the fact that the high lethality of ARDS is more associated to circulatory failure and less to hypoxemia. A ventilation strategy that ensures adequate gas exchange and at the same time causes as little additional stress as possible on the right heart would be optimal.

If the patient is eligible for the study according to the inclusion and exclusion criteria, an echocardiographic examination with 3D volumetric measurement of the right-sided heart cavities is performed. The conductance catheter will then be calibrated using this volumetric dataset. First, a conventional right heart catheterization is performed (conventional Swan-Ganz catheter), followed by the placement of the conductance catheter and the recording of a baseline. The "best PEEP" is then titrated by minimizing the "driving pressure" during volume-controlled ventilation as a descending sequence (from high PEEP to low PEEP). PV loops are recorded at each PEEP level. After determining the best PEEP level, the patient will be rotated to prone position. PV loops are recorded immediately after the rotation and within the following 45 minutes. The catheter is then removed. If the admixture of NO in the respiratory gas is indicated for medical reasons, the PV loops are recorded before and after the start of the admixture.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Invasive mechanical ventilation and clinical indication for prone positioning (e.g. ARDS)
* No contraindications for right heart catheterization or conductance catheterization
* The written consent of the patient or his legal guardian

Exclusion Criteria:

* No written consent
* contraindications for right heart catheterization or conductance catheterization
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study poulation consists of patients which require invasive ventilation as a result of a pulmonary disease and have a clinical need for prone positioning.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-11-04 (Estimated); Study Completion 2024-11-04 (Estimated)

PRIMARY OUTCOMES:
Changes in right ventricular pressure and volume and derived functional parameters caused by positive endexspiratory pressure | 15 minutes at each PEEP-Level
Changes in right ventricular pressure and volume and derived functional parameters caused by prone positioning | 1, 5, 10, 15, 20, 25, 35 and 45 minutes after rotation
Changes in right ventricular pressure and volume and derived functional parameters caused inhalation of NO | 10 minutes after start of NO-Administration

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Justus Liebig University Giessen, Universities of Giessen and Marburg Lung Center (UGMLC), German Center for Lung Research (DZL), Giessen, Hesse, Germany